CLINICAL TRIAL: NCT06302491
Title: A Study of Safety and Efficiency of AND017 in Patients With Transfusion Dependent and Non-transfusion Dependent β-thalassemia
Brief Title: A Study of Safety and Efficiency of AND017 in Patients With β-thalassemia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Kind Pharmaceuticals LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AND017-BTH-205
Record Dates: First submitted 2023-03-22; First posted 2024-03-08 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: β -Thalassemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- AND017 capsules 8 mg (Experimental)
  Interventions: Drug: AND017 capsules
- AND017 capsules 12 mg (Experimental)
  Interventions: Drug: AND017 capsules
- AND017 capsules 16 mg (Experimental)
  Interventions: Drug: AND017 capsules
- AND017 Placebo capsules (Placebo Comparator)
  Interventions: Drug: AND017 Placebo

INTERVENTIONS:
Drug: AND017 capsules — Administer AND017 capsules once per day (QD)
  Arms: AND017 capsules 12 mg; AND017 capsules 16 mg; AND017 capsules 8 mg
Drug: AND017 Placebo — Administer AND017 matching placebo capsules once per day (QD)
  Arms: AND017 Placebo capsules

SUMMARY:
This is a phase II, randomized, double-blinded, placebo-controlled study to treat patients with transfusion-dependent and non-transfusion dependent β -thalassemia with AND017 and optimal supportive care, including blood transfusion and iron removal, based on the clinician's judgment and practice.

ELIGIBILITY:
Inclusion Criteria:

1. Documented diagnosis of β-thalassemia or hemoglobin E/β-thalassemia, HbS/ β-thalassemia (β-thalassemia with α-bead mutation and/or multiplication is not allowed).
2. TDT subjects: receive regular blood transfusions, defined as 6-20 RBC units (including threshold) in the 24 weeks prior to screening assessment, and no transfusion-free period of ≥ 5 weeks during this period.
3. NTDT cohort: having transfused <6 RBC units in the 24 weeks prior to the screening assessment, no regular transfusion schedule, and no transfusion for 4 weeks prior to the screening assessment.
4. Subject transfusion records should be obtained within 24 weeks prior to the screening assessment, containing the date of transfusion, transfused RBC units, and pre-transfusion hemoglobin values.
5. ECOG score 0-1.
6. NTDT subjects with Hb ≤ 10.0 g/dL at screening test and one follow-up test (two tests more than one week apart) and difference in values between the two tests ≤ 1.0 g/dL.
7. Adequate liver function: Total bilirubin < 1.5 x upper limit of normal (ULN) (subjects with Gilbert syndrome, i.e., unconjugated hyperbilirubinemia, have a total bilirubin < 3 x ULN), aspartate aminotransferase

Exclusion Criteria:

1. Other causes of anemia (e.g., hemolytic anemia, history of pure red blood cell aplastic anemia, myelodysplastic syndrome, or multiple myeloma)
2. Presence of active infection or inflammatory disease requiring systemic anti-infective therapy, including concomitant autoimmune diseases with inflammatory symptoms (e.g. generalized erythema, ankylosing spondylitis, rheumatoid arthritis, psoriatic arthritis, dry syndrome, etc.)
3. Complicated retinal neovascularization requiring treatment (diabetic proliferative retinopathy, age-related exudative macular degeneration, retinal vein occlusion, macular edema, etc.)
4. Inability to take oral medications, conditions with a history of gastrectomy/bowel resection that may have an effect on the absorption of gastrointestinal medications (excluding gastric polyps or colonic polypectomy), or gastroparesis that remains symptomatic on current therapy
5. Clinically significant bleeding (requiring emergency blood transfusion within 12 h or a decrease in hemoglobin ≥ 2 g/dL within one week) within 4 weeks prior to the first dose, or a tendency to bleed or risk of bleeding that has not been medically or surgically corrected
6. Uncontrolled hypertension, defined as a diastolic blood pressure value >95 mmHg or a systolic blood pressure >160 mmHg on 2 or more of 3 repeated blood pressure tests (each at least 5 minutes apart) during the screening period
7. Complicated congestive heart failure (New York Heart Association [NYHA] class III or higher).
8. history of stroke, transient ischemic attack (TIA), myocardial infarction, thromboembolic event (deep vein thrombosis, DVT), pulmonary embolism, or pulmonary infarction within 24 weeks prior to screening evaluation
9. history of significant coagulation abnormalities, or platelet count >600 x 109/L or <80 x 109/L
10. History of epilepsy or any past seizures.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2024-05-27 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Evaluate the safety and tolerability of different oral doses of AND017 in the treatment of β-thalassemia subjects | From baseline to Week 24 or End of Treatment if discontinue early
  Evaluate the safety and tolerability of different oral doses of AND017 in the treatment of β-thalassemia subjects by AE rate by CTCAE 5.0

SECONDARY OUTCOMES:
Change in mean Hb levels relative to baseline at weeks 8-12 and week 20-24 post-treatment compared to baseline (mean Hb values during the 4 weeks prior to the first dose). | Baseline, Week 8-12, Week 20-24
  For NTDT cohort, evaluation of the effect of AND017+BSC on Hb levels.
The level of Hb and the change from baseline at each visit throughout the treatment period. | From baseline to Week1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 14, 16, 18, 20, 22, 24
  For NTDT cohort, evaluation of the effect of AND017+BSC on Hb levels.
Proportion of patients with mean Hb elevation ≥1.0 g/dL from baseline to weeks 8-12 after dosing. | Baseline, Week 8-12
  For NTDT cohort, evaluation of the effect of AND017+BSC on Hb levels.
Levels of and changes from baseline in red blood cell count throughout the treatment period | From baseline to Week1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 14, 16, 18, 20, 22, 24
  For NTDT cohort, Evaluation of the effect of AND017+BSC on RBC count
Levels of and changes from baseline in reticulocyte count throughout the treatment period | From baseline to Week1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 14, 16, 18, 20, 22, 24
  For NTDT cohort, Evaluation of the effect of AND017+BSC on reticulocyte count
Levels of and changes from baseline in mean corpuscular volume (MCV) throughout the treatment period | From baseline to Week1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 14, 16, 18, 20, 22, 24
  For NTDT cohort, Evaluation of the effect of AND017+BSC on the MCV
Levels of and changes from baseline in mean corpuscular hemoglobin (MCH) throughout the treatment period | From baseline to Week1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 14, 16, 18, 20, 22, 24
  For NTDT cohort, Evaluation of the effect of AND017+BSC on MCH
Levels of and changes from baseline in mean corpuscular hemoglobin concentration (MCHC) throughout the treatment period | From baseline to Week1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 14, 16, 18, 20, 22, 24
  For NTDT cohort, Evaluation of the effect of AND017+BSC on MCHC
Throughout the treatment period, changes in the levels and relative baseline of transferrin will be assessed. | From baseline to Week 4, 8, 12, 16, 20, 24
  For NTDT cohort, evaluation of the effect of AND017+BSC on transferrin level
Throughout the treatment period, changes in the levels and relative baseline of transferrin saturation (TSAT) will be assessed. | From baseline to Week 4, 8, 12, 16, 20, 24
  For NTDT cohort, evaluation of the effect of AND017+BSC on TSAT.
Throughout the treatment period, changes in the levels and relative baseline of ferritin will be assessed. | From baseline to Week 4, 8, 12, 16, 20, 24
  For NTDT cohort, evaluation of the effect of AND017+BSC on ferritin
Throughout the treatment period, changes in the levels and relative baseline of serum iron level will be assessed. | From baseline to Week 4, 8, 12, 16, 20, 24
  For NTDT cohort, evaluation of the effect of AND017+BSC on serum iron level
Throughout the treatment period, changes in the levels and relative baseline of total iron binding capacity (TIBC) will be assessed. | From baseline to Week 4, 8, 12, 16, 20, 24
  For NTDT cohort, evaluation of the effect of AND017+BSC on TIBC
Change in transfusion load (units transfused) at 12-24 weeks post-dose compared to baseline (12 weeks to W0 before first dose). | Baseline, Week 20-24, or End of Treatment if discontinue early
  For TDT cohort, evaluate changes in mean transfusion load by AND017+BSC at 12 to 24 weeks after dosing
Change in number of transfusions at 12-24 weeks post-dose compared to baseline (12 weeks to W0 before first dose). | Baseline and Week 20-24
  For TDT cohort, evaluate changes in mean transfusion load by AND017+BSC at 12 to 24 weeks after dosing
Proportion of subjects with ≥33% reduction in transfusion load (transfusion units) relative to baseline (12 weeks prior to first dose to W0) from baseline to any consecutive 12-week period after dosing. | Baseline, Week 0-12, 2-14, 4-16, 6-18, 8-20, 10-22, and 12-24
  For TDT cohort, proportion of subjects with ≥33% reduction in transfusion load (transfusion units) relative to baseline (12 weeks prior to first dose to W0) from baseline to any consecutive 12-week period after dosing.
Duration (days) of maintenance below this transfusion dose after a 33% reduction in transfusion load from baseline has been achieved. | From baseline to Week 24 or End of Treatment if discontinue early
  For TDT cohort, duration (days) of maintenance below this transfusion dose after a 33% reduction in transfusion load from baseline has been achieved.

CONTACTS AND LOCATIONS:
Overall Officials: Yusha Zhu, MD, PhD, Study Director — Kind Pharmaceuticals LLC
Locations (5):
- China (5):
  - Nanfang Hospital Southern Medical University, Guangzhou, Guangdong
  - Maoming People's Hospital, Maoming, Guangdong
  - Liuzhou People's Hospital, Liuchow, Guangxi
  - Guangxi Medical University No.1 Affiliated Hospital, Nanning, Guangxi
  - Hainan General Hospital, Haikou, Hainan